CLINICAL TRIAL: NCT03522558
Title: Medical Nutrition Therapy for Medically Complex Infants in the Pediatric Outpatient Setting. A Quality Improvement Project
Brief Title: Medical Nutrition Therapy for Medically Complex Infants in the Pediatric Outpatient Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Candice Rachel Poland, Registered Dietitian, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-18-0276
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Growth Failure in Medically Complex Infants; Growth Failure; Malnutrition in Medically Complex Infants; Malnutrition; Nutrition in Medically Complex Infants; Nutrition; Nutrition Disorder, Infant
MeSH Terms: conditions — Failure to Thrive; Malnutrition; Infant Nutrition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Medical Nutrition Therapy (Experimental): Standardized Medical Nutrition Therapy will include nutrition assessment provided by a registered dietitian (RD) at initial clinic visit or first Well Child Check (WCC) and regularly scheduled nutrition follow-up at each WCC visit thereafter.
  Interventions: Behavioral: Standardized Medical Nutrition Therapy
- Usual Care (Active Comparator): At the primary care provider's discretion, a nutrition consult can be requested for the RD to perform nutrition assessment or discuss the patient's plan without full nutrition assessment, as is current practice. Currently in the Neonatal High-Risk Clinic (NHRC) and High Risk Children's Clinic (HRCC) at UTHealth, providers consult the RD as deemed appropriate with no established criteria for when to include the RD in patient care. Usual care will not be modified by the study protocol.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Standardized Medical Nutrition Therapy — Standardized Medical Nutrition Therapy will include nutrition assessment provided by a registered dietitian (RD) at initial clinic visit or first Well Child Check (WCC) and regularly scheduled nutrition follow-up at each WCC visit thereafter.
  Arms: Standardized Medical Nutrition Therapy
Behavioral: Usual Care — At the primary care provider's discretion, a nutrition consult can be requested for the RD to perform nutrition assessment or discuss the patient's plan without full nutrition assessment, as is current practice. Currently in the Neonatal High-Risk Clinic (NHRC) and High Risk Children's Clinic (HRCC) at UTHealth, providers consult the RD as deemed appropriate with no established criteria for when to include the RD in patient care. Usual care will not be modified by the study protocol.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to compare standardized nutrition therapy provided by a registered dietitian (RD) at regularly scheduled intervals to usual care in terms of the ability to improve growth parameters in medically complex infants in the pediatric outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted between July, 2018 and June, 2019 to the Neonatal High-Risk Clinic (NHRC) and High Risk Children's Clinic (HRCC) at UT Health from a neonatal intensive care unit (NICU)

Exclusion Criteria:

* short bowel syndrome,
* requiring parenteral nutrition (PN)
* active cancer

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a 20% improvement in growth velocity at 1 year corrected gestational age (CGA) | 4 months corrected gestational age (CGA)
Number of participants with a 20% improvement in growth velocity at 1 year corrected gestational age (CGA) | 8 months corrected gestational age (CGA)
Number of participants with a 20% improvement in growth velocity at 1 year corrected gestational age (CGA) | 12 months corrected gestational age (CGA)
Number of participants with a 20% improvement in growth velocity at 1 year corrected gestational age (CGA) | 1 year corrected gestational age (CGA)

SECONDARY OUTCOMES:
Number of participants with growth failure | 1 year corrected gestational age (CGA)
  Growth failure ("Failure to Thrive") is defined as crossing 2 growth percentiles in a downward trajectory in the first year of life per child.
Number of participants who are malnourished | 1 year corrected gestational age (CGA)
  The Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition (AND/ASPEN) criteria are used for diagnosing pediatric malnutrition.
Severity of malnutrition as assessed by the AND/ASPEN criteria | 1 year corrected gestational age (CGA)
Number of emergency department visits | 1 year corrected gestational age (CGA)
Number of hospitalizations | 1 year corrected gestational age (CGA)
Length of stay | about 3 to 7 days
  number of hospital days

CONTACTS AND LOCATIONS:
Overall Officials: Candice R Poland, MS, RD, LD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States